CLINICAL TRIAL: NCT02470429
Title: Evaluation of Clinical Outcomes Following the Use of SYSTANE® HYDRATION in Subjects With Dry Eye
Brief Title: Evaluation of Clinical Outcomes After the Use of SYSTANE® HYDRATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXK947-P001
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYSTANE HYDRATION (Experimental): SYSTANE HYDRATION lubricant eye drops, 1 drop 4 times per day (QID) in each eye for 42 days
  Interventions: Device: SYSTANE HYDRATION lubricant eye drops; Drug: 0.9% saline eye drops
- Hyabak 0.15% (Active Comparator): Hyabak 0.15% eye drops, 1 drop 4 times per day (QID) in each eye for 42 days
  Interventions: Device: Hyabak 0.15% eye drops; Drug: 0.9% saline eye drops

INTERVENTIONS:
Device: SYSTANE HYDRATION lubricant eye drops — Preserved with POLYQUAD (polidronium chloride) 0.001%
  Other Names: SYSTANE® HYDRATION
  Arms: SYSTANE HYDRATION
Device: Hyabak 0.15% eye drops — Preservative-free
  Other Names: Hyabak 0.15%
  Arms: Hyabak 0.15%
Drug: 0.9% saline eye drops — Preservative-free, one drop 4 times a day in each eye (run-in period)

SUMMARY:
The purpose of this study is to compare SYSTANE® HYDRATION to Hyabak 0.15% based on total ocular surface staining scores (TOSS) at Day 42.

DETAILED DESCRIPTION:
Subjects will first be dispensed preservative-free 0.9% saline eye drops (saline eye drops) to be used during the Run-in phase between Screening Visit and Day 0 (Visit 1). Subjects who qualify will be randomized in a 1:1 manner to receive either treatment with SYSTANE® HYDRATION Lubricant Eye Drops or Hyabak 0.15% Eye Drops.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to attend all study visits;
* Use of non-BAK (Benzalkonium Chloride) artificial tears at least once a day, for at least 3 months prior to Screening Visit;
* Diagnosis of Dry Eye (by a health care professional) for at least 3 months prior to Screening Visit;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential who are pregnant or breast feeding;
* Any hypersensitivity to the use of the study products or an allergy to any ingredient(s) contained within study products;
* Ocular abnormalities in either eye that could adversely affect the safety or efficacy outcome;
* Active ocular infection (bacterial, viral, or fungal) or active inflammation not associated with dry eye;
* Use of chronic systemic medications: (prescription, over the counter, vitamins/supplements) on a stable dose for less than 30 days prior to Screening Visit, or any anticipated change in dosing regimen during the course of the study;
* History of ocular or intraocular surgery or serious ocular trauma in either eye within 6 months prior to Screening Visit;
* Any medical condition (systemic or ophthalmic) that may, in the opinion of the Investigator, preclude the safe administration of study products or safe participation in the study;
* Use of any topical ocular over-the-counter or prescribed medications in either eye (with the exception of artificial tears/gels/ lubricants) 2 weeks prior to Screening Visit;
* Contact lens use within 2 weeks prior to Screening Visit and unwilling to avoid contact lens use during the course of the study;
* Unwilling to avoid the use of additional artificial tears (other than the study products) throughout the study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Trial Leader, Global Development Operations, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 study centers located in Germany, 3 study centers located in France, 2 study centers located in the UK, and 2 study centers located in Spain.
Pre-assignment Details: Of the 114 enrolled, 15 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (99).
Period: Overall Study
Arm/Group | SYSTANE HYDRATION | Hyabak 0.15%
Started | 50 | 49
Completed | 48 | 49
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who were exposed to study drug (including the run-in therapy) (Safety Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | SYSTANE HYDRATION | Hyabak 0.15% | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (12.29) | 56.7 (14.29) | 59.2 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 79
  Male | 9 | 11 | 20
Total Ocular Surface Staining (TOSS) Score [Mean (Standard Deviation); unit: units on a scale] — The TOSS score is a cumulative cornea and conjunctival staining score. After instilling ophthalmic dye in the eye, the investigator graded 3 areas of the ocular surface for dryness on a scale from 0 to 5, where 0=Absent and 5=Severe. The 3 scores were summed for a resultant overall 0-15 score. Population: This analysis population includes all subjects who received at least 1 dose of the randomized study drug (Intent-to-Treat (ITT) Analysis Set).
  units on a scale | 5.26 (1.411) | 4.98 (1.090) | 5.12 (1.264)
IDEEL Treatment Score [Mean (Standard Deviation); unit: units on a scale] — The IDEEL (Impact of dry eye on everyday life) is 10-question patient-reported outcome questionnaire that assesses the subject's general satisfaction with treatment use (Treatment Effectiveness and Treatment Inconvenience). A resultant overall 0-100 treatment satisfaction score was calculated separately for Treatment Effectiveness and Treatment Inconvenience, with higher scores indicating greater satisfaction and less treatment-related bother. Population: ITT Analysis Set. Number Analyzed is the number of subjects with non-missing response.
  units on a scale
    Treatment Effectiveness: number analyzed (Participants) | 49 | 48 | 97
    Treatment Effectiveness | 52.04 (29.602) | 51.56 (28.641) | 51.80 (28.979)
    Treatment Inconvenience: number analyzed (Participants) | 49 | 48 | 97
    Treatment Inconvenience | 83.42 (17.749) | 81.90 (17.829) | 82.67 (17.712)
Tear Film Break-up Time (TFBUT) [Mean (Standard Deviation); unit: seconds] — TFBUT is defined as the time elapsed from the last blink until 1 or more dry spots appeared in the precorneal tear film. Population: ITT Analysis Set.
  seconds | 3.20 (2.010) | 3.58 (2.222) | 3.39 (2.115)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Ocular Surface Staining (TOSS) Score at Day 42
Description: The TOSS score is a cumulative cornea and conjunctival staining score. After instilling ophthalmic dye in the eye, the investigator graded 3 areas of the ocular surface for dryness on a scale from 0 to 5, where 0=Absent and 5=Severe. The 3 scores were summed for a resultant overall 0-15 score. A more negative change value indicates greater efficacy. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Day 42
Population: ITT Analysis Set. Number Analyzed is the number of subjects with non-missing response.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SYSTANE HYDRATION | Hyabak 0.15%
Number analyzed (Participants) | 48 | 49
units on a scale | -1.16 (0.24) | -0.92 (0.23)

2. Secondary Outcome: Change From Baseline in IDEEL Treatment Effectiveness Score at Day 42
Description: The IDEEL is 10-question patient-reported outcome questionnaire that assesses the subject's general satisfaction with treatment use. A resultant overall 0-100 satisfaction score was calculated, with a higher score indicating greater satisfaction and less treatment-related bother.
Time Frame: Baseline (Day 0), Day 42
Population: ITT Analysis Set. Number Analyzed is the number of subjects with non-missing response.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SYSTANE HYDRATION | Hyabak 0.15%
Number analyzed (Participants) | 47 | 48
units on a scale | 9.62 (3.19) | 12.80 (3.17)

3. Secondary Outcome: Change From Baseline in IDEEL Treatment Inconvenience Score at Day 42
Description: as for outcome 2
Time Frame: Baseline (Day 0), Day 42
Population: ITT Analysis Set. Number Analyzed is the number of subjects with non-missing response.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SYSTANE HYDRATION | Hyabak 0.15%
Number analyzed (Participants) | 47 | 47
units on a scale | -10.32 (2.22) | 2.24 (2.22)

4. Secondary Outcome: Change From Baseline in Tear Film Break-up Time (TFBUT) at Day 42
Description: TFBUT is defined as the time elapsed from the last blink until 1 or more dry spots appeared in the precorneal tear film. A longer tear film break-up time indicates a more stable tear film and may lead to improvement in dry eye symptoms. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Day 42
Population: ITT Analysis Set. Number Analyzed is the number of subjects with non-missing response.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | SYSTANE HYDRATION | Hyabak 0.15%
Number analyzed (Participants) | 48 | 49
seconds | 0.39 (0.38) | 0.68 (0.37)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 63 days). AEs are reported as pretreatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence in a subject who was administered an investigational product regardless of whether or not the event had a causal relationship with the treatment. AEs were obtained through volunteered and elicited comments from subjects and through observations by the Investigator.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to the initiation of study treatment
- SYSTANE HYDRATION: All subjects treated with SYSTANE HYDRATION lubricant eye drops
- Hyabak 0.15%: All subjects treated with Hyabak 0.15% eye drops
Arm/Group | Pretreatment | SYSTANE HYDRATION | Hyabak 0.15%
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/114 | 1/50 | 1/49
Other Adverse Events (participants affected / at risk) | 2/114 | 12/50 | 6/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=114) | SYSTANE HYDRATION (N=50) | Hyabak 0.15% (N=49)
Intervertebral disc operation (Surgical and medical procedures) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=114) | SYSTANE HYDRATION (N=50) | Hyabak 0.15% (N=49)
Eye irritation (Eye disorders) | 0 | 5 | 3
Vision blurred (Eye disorders) | 0 | 5 | 1
Nasopharyngitis (Infections and infestations) | 1 | 5 | 1
Headache (Nervous system disorders) | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.